CLINICAL TRIAL: NCT00005650
Title: Genetic Study of Patients With Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of North Carolina (Other)
Other Study IDs: NCRR-M01RR00046-1395; UNCCH-GCRC-1395
Record Dates: First submitted 2000-05-02; First posted 2000-05-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: cardiovascular and respiratory diseases; genetic diseases and dysmorphic syndromes; primary ciliary dyskinesia; rare disease
MeSH Terms: conditions — Ciliary Motility Disorders; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
OBJECTIVES:

I. Characterize the clinical presentation of patients with primary ciliary dyskinesia.

II. Identify the genetic mutations associated with this disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Participants undergo a scrape biopsy acquisition of nasal cells for ciliary studies, a chest radiograph, sinus radiographs, lung function tests, sputum cultures, nitric oxide measurement, and an ear, nose and throat evaluation to screen for primary ciliary dyskinesia (PCD). Blood collection and/or a buccal scrape is also performed for genetic studies.

Genetic studies include molecular linkage analyses, genetic mapping, and gene mutation identification based on large deletions. Microsatellite markers are used to identify polymorphism.

Genetic counseling is provided to all participants.

ELIGIBILITY:
* Histologically or cytologically confirmed primary ciliary dyskinesia (PCD)
* Family members of patients with PCD

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: Peadar G. Noone, Study Chair — University of North Carolina
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States